CLINICAL TRIAL: NCT05154773
Title: Increasing Live Donor Kidney Transplantation Through Video-based Education and Mobile Communication
Acronym: KidneyTIME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Liise Kayler, Primary Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00005449
Record Dates: First submitted 2021-11-16; First posted 2021-12-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: End-stage Renal Disease; Chronic Kidney Diseases
Keywords: Kidney transplant access; living kidney donation; education; web-based intervention; randomized controlled trial
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KidneyTIME (Experimental): KidneyTIME is a self-directed digital intervention. It contains 26 animated videos, each 1-3 minutes in length, designed to address knowledge gaps and concerns about kidney transplantation and living donation that were identified in literature reviews, formative research, and video development studies as critical for optimal prospective kidney recipient and donor participation in LDKT. We chose 6 videos from the entire series to be delivered sequentially for a total duration of 13 minutes. After completing the proscribed videos and an immediate-post exposure survey, everyone then received a link to access all 26 videos centralized on a website where the videos were activated for sharing through various modalities, including text, email, Facebook, and Twitter. The website could be accessed using this link from any electronic device throughout the study. Prompts to use the intervention were sent once a week for 3 weeks and then monthly for 12 months.
  Interventions: Behavioral: Kidney donation and transplant information made easy
- Usual Care (No Intervention): Routine educational materials from non-study sources through usual Transplant Center protocols including booklets, nurse communications, and the usual care video, a nurse-narrated power-point presentation outlining recipient and donor evaluation, surgery, and recovery processes and outcomes.

INTERVENTIONS:
Behavioral: Kidney donation and transplant information made easy — Same as arm description
  Other Names: KidneyTIME
  Arms: KidneyTIME

SUMMARY:
The study is a- 2-arm randomized controlled trial among patients presenting for kidney transplant evaluation at a single transplant center to compare the effects of a patient-based self-learning and outreach intervention about living-donor kidney transplantation (KidneyTIME) versus usual care for living-donor kidney transplant knowledge, concerns, readiness, access behaviors, and living-donor inquiries over 12 months follow-up. Following consent and baseline assessment, participants were randomized, stratified by self-reported race, with equal allocation to 2 treatment arms: the KidneyTIME intervention and usual care.

DETAILED DESCRIPTION:
Over a 2.5 year period we will conduct a 2-arm parallel randomized trial among patients presenting for kidney transplant evaluation at a single transplant center to compare the effects of KidneyTIME versus usual care for KTX access over 12 months of intervention use and follow-up.

Participants will be recruited from the Transplant program at Erie County Medical Center, a safety-net hospital in Buffalo, New York. Each week, electronic records will be accessed to identify potential participants who had been referred to the transplant center for a kidney transplant, are aged 18 years and older, speak English, have internet access, and signed electronic consent as well as provided a text or email address. We will excude patients previously exposed to any component of the intervention.

Each potential participant will be sent an electronic invitation from the principal investigator (a transplant surgeon). This message will briefly described the study and include a personal link to an online consent form describing study procedures and potential risks. A stakeholder Advisory Council, whose members include patients and care partners, will review and provide ongoing feedback on the recruitment and retention plan.

The entire study and the progress tracker will be hosted on Alchemer. Those who sign electronic consent to participate will be automatically guided to a baseline sociodemographic survey (T0). Upon completion, computer-generated randomization will stratify participants by self-reported race (Black versus Other), with equal allocation to 2 treatment arms: the KidneyTIME intervention and usual care. Condition assignment of each participant will be concealed from transplant providers, but participants will become aware of their treatment assignment one they access the study educational content.

KidneyTIME is a self-directed digital intervention. It contains 26 animated videos, each 1-3 minutes in length, designed to address knowledge gaps and concerns about kidney transplantation and living donation that were identified in literature reviews, formative research, and video development studies as critical for optimal prospective kidney recipient and donor participation in LDKT. All components of the intervention were developed through a user-centered design approach by involving kidney failure patients and social network members, to improve usability and increase the likelihood of adoption.

In the intervention arm, we chose 6 videos from the entire series to be delivered sequentially for a total duration of 13 minutes. The first video sets the stage for the intervention and introduces the viewer to an overview of LDKT. The next 5 videos address common misconceptions about live kidney donation: Video 1: LDKT introduction, Video 2: Donor eligibility, Video 3: Donor evaluation, Video 4: Kidney paired donation, Video 5: Donation Costs, Video 6: Donor lifestyle. After completing the proscribed videos and an immediate-post exposure survey, everyone then receives a link to access all 26 videos centralized on a website where the videos were activated for sharing through various modalities, including text, email, Facebook, and Twitter. The website can be accessed using this link from any electronic device throughout the study. Website use will be prompted by automated messages (email or SMS) that introduced videos that may interest users, provided the website link, and encouraged video viewing and sharing. Messages will be personalized with their name and provide researchers contact information. Prompts will be sent monthly for 12 months.

Control participants will receive the transplant program's 13-minute usual care video, a nurse-narrated power-point-based video outlining recipient evaluation, surgery, recovery processes and outcomes while highlighting the option of LDKT. This condition was active since it intended to aid kidney transplant access. It was utilized to offer participants education with perceived benefit and encourage further study participation.

All participants routinely receive educational materials from non-study sources through usual Transplant Center protocols including written materials, nurse communications, and the usual care video shown on a clinic computer during transplant evaluation. Therefore control participants viewed the usual care video twice.

After completing the proscribed video education, all participants will be invited to fill out serial surveys immediately (T1) and 1 month (T2), 6 months (T3), and 12-months (T4) post-baseline. Participants will receive up to 6 reminders (5 automatic and 1 personalized) to complete surveys. At study conclusion, intervention participants will be invited to an exit interview and controls will be offered access to the intervention website. All participants will receive up to $125 for completing study milestones (4 surveys and an exit interview).

ELIGIBILITY:
Inclusion Criteria:

* referred to the transplant center for a kidney transplant
* aged 18 years and older
* speaks English
* has access to the internet

Exclusion Criteria:

* Previously exposed to any component of the intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Living Donor Inquiry | 12 months
  Living donor inquiry to the transplant center on behalf of the participant by telephone, email, or mail within 12 months from enrollment. Each inquiry is captured for all patients as a discrete field in the electronic medical record within 12 months from enrollment. An inquiry includes any request for information or evaluation to be a living kidney donor. in which the recipient is specified.

SECONDARY OUTCOMES:
LDKT Knowledge scale | immediately post baseline, 1 month, 6 month, and 12 months
  Developed specifically for this study as a measure of patients' knowledge about LDKT as delivered in the intervention condition. In this 12-item true-false questionnaire, total scores range from 0-12 with higher scores indicating greater LDKT-related knowledge. The scale captured different dimensions of knowledge including donor eligibility criteria, clinical outcomes, costs of the donation procedure, donor diet and medications, donor priority for transplant, and kidney paired donation.
LDKT Concerns Scale | immediately post baseline, 1 month, 6 month, and 12 months
  Developed specifically for this study as a measure of patients' concerns about LDKT. Questions were drawn from existing measures in the literature. We created a 6-items scale that captured concerns about LDKT including donation costs, evaluation process, function with a single kidney, poor outcome, and surgical risk as well as one question about access to deceased-donor kidney transplantation. Items are rated on a scale of 1 to 4. Higher scores indicate greater concerns about live kidney donation.
LDKT Readiness | immediately post baseline, 1 month, 6 month, and 12 months
  A measure of one's readiness for living-donor kidney transplantation. This 1-item scale measures the degree to which a person is ready for LDKT and is adapted from existing measures in the literature. Response options correspond to 5 stages of change based on the Transtheoretical Model and Stages of Change and are rated on a scale of 1 to 5, with higher scores indicating greater readiness.
LDKT action behaviors | immediately post baseline, 1 month, 6 month, and 12 months
  A measure of ongoing progress toward living donor kidney transplantation or waitlisting. To assess LDKT action behaviors patients will be asked whether they had done any of 11 transplant-related behaviors adapted from existing measures in the literature. Patients who indicated they had done the action will counted and scores will range from 0 to 11.

OTHER OUTCOMES:
Time to waiting-list placement | 12 months
  The first time from evaluation to active placement on the kidney transplant waiting list will assessed via medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Liise Kayler, MD, Principal Investigator — University at Buffalo
Locations (1):
- Erie County Medical Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make all data available upon request.
Supporting Information: CSR
Time Frame: The deidentified participant data and data dictionary data set will be made available upon request. The dataset will be archived for at least 10 years after publication.
Access Criteria: Researcher meets University at Buffalo IRB guidelines for data sharing. Request to the PI team at our institution for any valid scientific purpose and after publication